CLINICAL TRIAL: NCT00350103
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Trial to Assess the Efficacy and Safety of 400mg/Day Lacosamide in Subjects With Painful Distal Diabetic Neuropathy Using Two Different Titration Schemes
Brief Title: A Trial to Assess the Efficacy and Safety of 400mg/Day Lacosamide in Subjects With Painful Diabetic Neuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Collaborators: SCHWARZ BIOSCIENCES GmbH - Part of UCB Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP0874; 2005-005788-27 (EudraCT Number)
Record Dates: First submitted 2006-07-06; First posted 2006-07-10 (Estimated); Results first posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2023-09

CONDITIONS: Painful Diabetic Neuropathy
Keywords: Painful Diabetic Neuropathy; Lacosamide
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Lacosamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lacosamide Standard Titration (ST) (Experimental): Subjects had their dose titrated from 100 mg/day to 400 mg/day at weekly intervals of 100 mg. Subjects in this treatment group reach their target dose of 400 mg/day 3 weeks after Visit 2. All subjects completing the Titration Phase enter a 12-week Maintenance Phase.
  Interventions: Drug: SPM 929
- Lacosamide Fast Titration (FT) (Experimental): Subjects receive 200 mg/day LCM for the first 3 days, 300 mg/day for the next 4 days, and reach their target dose of 400 mg/day after 1 week. They undergo sham titration for the remaining 3 weeks of the Titration Phase. All subjects completing the Titration Phase enter a 12-week Maintenance Phase.
  Interventions: Drug: SPM 929
- Placebo (Placebo Comparator): Subjects underwent sham titration for the entire Titration Phase. All subjects completing the Titration Phase enter a 12-week Maintenance Phase
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPM 929 — * Pharmaceutical form: Immediate release film-coated tablets
  * Concentration: 50mg/ 100mg
  * Route of administration: Oral use
  Other Names: Lacosamide
  Arms: Lacosamide Fast Titration (FT); Lacosamide Standard Titration (ST)
Drug: Placebo — * Pharmaceutical form: Immediate release film-coated tablets
  * Route of administration: Oral use
  Arms: Placebo

SUMMARY:
The purpose of this trial is to assess whether 400mg/day of lacosamide is effective in reducing pain caused by distal diabetic neuropathy. Two dose-escalation schemes for lacosamide will be used to further determine the efficacy of the "standard" scheme and to evaluate the efficacy and safety of a more rapid titration scheme. Subjects will be randomly assigned to one of three treatment groups. Subjects in two of the groups will receive lacosamide at a dose of 400mg/day, but different dose-escalation schemes will be used to reach this final dose. The third group of subjects will receive a placebo. Subjects will have a 2 in 3 (66 %) chance of getting lacosamide.

The maximum lacosamide dose in this trial will be 400mg/day. The maximum treatment duration will be 18 weeks, including a two-week Pre-Treatment Phase and a 12 weeks period on a stable dose of lacosamide or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subject has had symptoms of painful diabetic neuropathy for at least 6 months and has a diagnosis of diabetes mellitus (Type I or Type II).

Exclusion Criteria:

* Subject has previously participated in this trial or subject has previously been assigned to treatment in a trial of the drug under investigation in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 551 (Actual)
Dates: Start 2006-06-30 (Actual); Primary Completion 2007-06-29 (Actual); Study Completion 2007-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (1):
- Monheim, Germany

REFERENCES:
- [Result] Bainbridge J, De Backer M, Eckhardt K, Tennigkeit F, Bongardt S, Sen D, Werhahn KJ, Shaibani A, Faught E. Safety and tolerability of lacosamide monotherapy in the elderly: A subgroup analysis from lacosamide trials in diabetic neuropathic pain. Epilepsia Open. 2017 Sep 11;2(4):415-423. doi: 10.1002/epi4.12079. eCollection 2017 Dec. PMID 29588972
- See also: Clinical Study Summary on UCB.com — https://www.ucb.com/website/_up/ucb_com_patients/documents/SP874_CSS_20080610.pdf
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in June 2006 and concluded in June 2007.
Pre-assignment Details: Participant Flow refers to the Randomized Set. The 16-week Treatment Phase consisted of 4-week Titration Phase and 12-week Maintenance Phase.
Groups:
- Lacosamide Standard Titration (ST): Subjects had their dose titrated from 100 mg/day to 400 mg/day at weekly intervals of 100mg. Subjects in this treatment group reach their target dose of 400 mg/day 3 weeks after Visit 2. All subjects completing the Titration Phase enter a 12-week Maintenance Phase.
Period: Overall Study
Arm/Group | Placebo | Lacosamide Fast Titration (FT) | Lacosamide Standard Titration (ST)
Started | 179 | 190 | 182
Entered Titration Phase (Received at least 1 dose of study medication (Safety Set)) | 179 | 189 | 181
Completed Titration Phase | 162 | 164 | 165
Entered Maintenance Phase | 162 | 163 | 164
Completed Maintenance Phase | 150 | 149 | 148
Completed | 149 | 148 | 146
Not Completed | 30 | 42 | 36
Not completed — Adverse Event | 12 | 29 | 17
Not completed — Lack of Efficacy | 5 | 1 | 3
Not completed — Withdrawal by Subject | 6 | 6 | 8
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Unsatisfactory Compliance | 2 | 2 | 1
Not completed — Investigator´s decision | 1 | 1 | 0
Not completed — Exclusion criteria met | 0 | 0 | 1
Not completed — Patient relocated | 0 | 0 | 1
Not completed — Need for prohibited medication | 1 | 0 | 0
Not completed — Personal reasons | 0 | 0 | 1
Not completed — Patient stopped feeling pain | 1 | 0 | 0
Not completed — PR greater than 250ms | 0 | 0 | 1
Not completed — Wrong calculation of QT interval | 0 | 0 | 1
Not completed — Sponsor mistake | 1 | 0 | 0
Not completed — Randomization mistake | 0 | 1 | 1
Not completed — Sponsor´s decision | 0 | 1 | 0
Not completed — Lost, Reason unknown | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Randomized Set which included all enrolled participants who were randomized to a specific treatment arm.
Groups:
- Lacosamide FT: Subjects receive 200 mg/day LCM for the first 3 days, 300 mg/day for the next 4 days, and reach their target dose of 400 mg/day after 1 week. They undergo sham titration for the remaining 3 weeks of the Titration Phase. All subjects completing the Titration Phase enter a 12-week Maintenance Phase.
- Lacosamide ST: Subjects had their dose titrated from 100 mg/day to 400 mg/day at weekly intervals of 100mg. Subjects in this treatment group reach their target dose of 400 mg/day 3 weeks after Visit 2. All subjects completing the Titration Phase enter a 12-week Maintenance Phase.
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST | Total Title
Number analyzed (Participants) | 179 | 190 | 182 | 551
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 142 | 147 | 134 | 423
  >=65 years | 37 | 43 | 48 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (9.45) | 58.0 (9.46) | 57.4 (10.14) | 57.3 (9.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 98 | 88 | 272
  Male | 93 | 92 | 94 | 279

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Daily Pain Score From Baseline Week to the Last 4 Weeks of the Maintenance Phase
Description: An 11-point Likert scale is used to assess the subject's average daily pain. This scale is completed by the subject twice daily (once in the morning and once in the evening). The subject rates his/her average pain over the last 12 hours, from 0 (no pain) to 10 (worst pain ever experienced). The daily pain score is defined as the average score of those collected in the morning and evening. The value reported below is calculated as a difference between the average of the last available 28 days of maintenance for participants completing the maintenance phase (or the last 28 days prior to discontinuation for participants who discontinued in the titration or maintenance phase) and the average of the Baseline week.
Time Frame: Last 4 weeks of Maintenance Phase, compared to the Baseline Week
Population: Only subjects with available data for subject's average daily pain scores are included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 177 | 188 | 177
units on a scale | -1.9 (2.20) | -2.2 (2.05) | -2.4 (2.08)
Statistical Analysis 1: Comparison: Placebo vs Lacosamide ST; Last Observation Carried Forward (LOCF) procedure was applied for missing daily diary entries between start of trial medication and Visit 8 or last intake of trial medication in the case of discontinuation during the Titration or Maintenance Phase; Test type: Superiority or Other; p = 0.0410, ANCOVA; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-0.88 to -0.02] — Estimated value is the difference of Least Square Means
Statistical Analysis 2: Comparison: Placebo vs Lacosamide FT; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2902, ANCOVA; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.65 to 0.20] — Estimated value is the difference of Least Square Means

2. Secondary Outcome: Time to Sustainable Pain Relief
Description: Time to sustainable pain relief was defined as the time from Baseline to the first day on which there was a ≥1-point improvement over Baseline in the Likert pain score for those subjects for whom there was also ≥30% reduction in average daily pain score over the last 28 days of the Maintenance Phase as compared to Baseline.
Time Frame: From start of trial medication intake (Week 0) up to the last 4 weeks of the Maintenance Phase
Population: Only subjects with available data for subject's average daily pain scores are included in the analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 177 | 188 | 177
days | 31.0 [11.0 to NA] — Upper confidence limits are not provided for the 95% CI of the median time to sustainable pain relief when there is no observed sustainable pain relief time for which the upper bound of the confidence interval for the Kaplan-Meier estimate is less than 0.5. | 11.0 [7.0 to 35.0] | 10.0 [6.0 to NA] — Upper confidence limits are not provided for the 95% CI of the median time to sustainable pain relief when there is no observed sustainable pain relief time for which the upper bound of the confidence interval for the Kaplan-Meier estimate is less than 0.5.

3. Secondary Outcome: Percentage of Subjects With >= 30% or >= 2-point Reduction of with-in Subject Change in Average Daily Pain Score From the Baseline Week to the Last 4 Weeks of the Maintenance Phase
Description: An 11-point Likert scale is used to assess the subject's average daily pain. This scale is completed by the subject twice daily (once in the morning and once in the evening). The subject rates his/her average pain over the last 12 hours, from 0 (no pain) to 10 (worst pain ever experienced). The daily pain score is defined as the average score of those collected in the morning and evening.
Time Frame: Baseline week, last 4 weeks of the Maintenance Phase
Population: Only subjects with available data for subject's average daily pain scores are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 177 | 188 | 177
percentage of participants | 50.3 | 56.4 | 55.4

4. Secondary Outcome: Within-subject Change in Average Daily Pain Score From the Baseline Week to Visit 3
Description: An 11-point Likert scale is used to assess the subject's average daily pain. This scale is completed by the subject twice daily (once in the morning and once in the evening). The subject rates his/her average pain over the last 12 hours, from 0 (no pain) to 10 (worst pain ever experienced). The daily pain score is defined as the average score of those collected in the morning and evening. A negative value indicates improvement from Baseline.
Time Frame: Baseline week, Visit 3
Population: Only subjects with available data for subject's average daily pain scores at the respective are included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 177 | 188 | 177
units on a scale | -0.5 (1.13) | -0.7 (1.07) | -0.7 (1.06)

5. Secondary Outcome: Within-subject Change in Average Daily Pain Score From the Baseline Week to Visit 4
Description: as for outcome 4
Time Frame: Baseline week, Visit 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 171 | 182 | 170
units on a scale | -0.9 (1.47) | -1.4 (1.63) | -1.3 (1.50)

6. Secondary Outcome: Within-subject Change in Average Daily Pain Score From the Baseline Week to Visit 5
Description: as for outcome 4
Time Frame: Baseline week, Visit 5
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 168 | 172 | 169
units on a scale | -1.3 (1.73) | -1.7 (1.87) | -1.8 (1.69)

7. Secondary Outcome: Within-subject Change in Average Daily Pain Score From the Baseline Week to Visit 6
Description: as for outcome 4
Time Frame: Baseline week, Visit 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 162 | 163 | 164
units on a scale | -1.9 (2.01) | -2.1 (2.08) | -2.2 (1.94)

8. Secondary Outcome: Within-subject Change in Average Daily Pain Score From the Baseline Week to Visit 7
Description: as for outcome 4
Time Frame: Baseline week, Visit 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 157 | 153 | 152
units on a scale | -2.2 (2.09) | -2.3 (2.03) | -2.5 (1.98)

9. Secondary Outcome: Within-subject Change in Average Daily Pain Score From the Baseline Week to Visit 8
Description: as for outcome 4
Time Frame: Baseline week, Visit 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 152 | 151 | 150
units on a scale | -2.2 (2.17) | -2.5 (2.07) | -2.6 (2.07)

10. Secondary Outcome: Within-subject Change in Average Daily Pain Score From the Baseline Week to the Titration Phase
Description: An 11-point Likert scale is used to assess the subject's average daily pain. This scale is completed by the subject twice daily (once in the morning and once in the evening). The subject rates his/her average pain over the last 12 hours, from 0 (no pain) to 10 (worst pain ever experienced). The daily pain score is defined as the average score of those collected in the morning and evening. A negative value indicates improvement from Baseline. The value reported below is calculated as a difference between the average of the titration phase and the average of the Baseline Week.
Time Frame: Titration Phase (4 weeks), compared to the Baseline Week
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 177 | 188 | 177
units on a scale | -1.0 (1.40) | -1.3 (1.47) | -1.4 (1.35)

11. Secondary Outcome: Within-subject Change in Average Daily Pain Score From the Baseline Week to the Maintenance Phase
Description: An 11-point Likert scale is used to assess the subject's average daily pain. This scale is completed by the subject twice daily (once in the morning and once in the evening). The subject rates his/her average pain over the last 12 hours, from 0 (no pain) to 10 (worst pain ever experienced). The daily pain score is defined as the average score of those collected in the morning and evening. A negative value indicates improvement from Baseline. The value reported below is calculated as a difference between the average of the maintenance phase and the average of the Baseline Week.
Time Frame: Maintenance Phase (12 weeks), compared to the Baseline Week
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 162 | 163 | 164
units on a scale | -2.1 (2.04) | -2.3 (1.98) | -2.3 (1.92)

12. Secondary Outcome: Within-subject Change in Average Daily Pain Score From the Baseline Week to the Treatment Phase
Description: An 11-point Likert scale is used to assess the subject's average daily pain. This scale is completed by the subject twice daily (once in the morning and once in the evening). The subject rates his/her average pain over the last 12 hours, from 0 (no pain) to 10 (worst pain ever experienced). The daily pain score is defined as the average score of those collected in the morning and evening. A negative value indicates improvement from Baseline. The value reported below is calculated as a difference between the average of the treatment phase and the average of the Baseline Week.
Time Frame: Treatment Phase (16 weeks), compared to the Baseline Week
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 177 | 188 | 177
units on a scale | -1.6 (1.83) | -1.9 (1.76) | -2.0 (1.72)

13. Secondary Outcome: Within-subject Change in Average Daily Pain Score From the Baseline Week to the Last 4 Weeks of Maintenance Phase
Description: An 11-point Likert scale is used to assess the subject's average daily pain. This scale is completed by the subject twice daily (once in the morning and once in the evening). The subject rates his/her average pain over the last 12 hours, from 0 (no pain) to 10 (worst pain ever experienced). The daily pain score is defined as the average score of those collected in the morning and evening. A negative value indicates improvement from Baseline. The value reported below is calculated as a difference between the average of the last available 28 days of maintenance for participants completing the maintenance phase (or the last 28 days prior to discontinuation for participants who discontinued in the titration or maintenance phase) and the average of the Baseline week.
Time Frame: Last 4 weeks of Maintenance Phase, compared to the Baseline Week
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 177 | 188 | 177
units on a scale | -1.9 (2.20) | -2.2 (2.05) | -2.4 (2.08)

14. Secondary Outcome: Within-subject Change From the Baseline Week to Visit 3 in Daily Perception of Pain Interference With Subject's Sleep
Description: An 11-point Likert scale was used to assess the subject's sleep. The subject rated how the pain had interfered with sleep over the past 12 hours, from 0 (no interference) to 10 (complete interference). A lower value on the scale indicates improvement in symptoms. A negative change value indicates improvement from Baseline. Baseline Week was defined as the average of pain interference scores at the last 7 days prior to Visit 2.
Time Frame: Baseline Week, Visit 3
Population: Only subjects with available data for subject's pain interference with subject's sleep at the respective are included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 177 | 186 | 176
units on a scale | -0.5 (1.27) | -0.7 (1.26) | -0.6 (1.35)

15. Secondary Outcome: Within-subject Change From the Baseline Week to Visit 4 in Daily Perception of Pain Interference With Subject's Sleep
Description: as for outcome 14
Time Frame: Baseline Week, Visit 4
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 171 | 180 | 169
units on a scale | -0.9 (1.72) | -1.3 (1.69) | -1.3 (1.83)

16. Secondary Outcome: Within-subject Change From the Baseline Week to Visit 5 in Daily Perception of Pain Interference With Subject's Sleep
Description: as for outcome 14
Time Frame: Baseline Week, Visit 5
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 168 | 170 | 168
units on a scale | -1.4 (1.87) | -1.7 (2.04) | -1.8 (2.01)

17. Secondary Outcome: Within-subject Change From the Baseline Week to Visit 6 in Daily Perception of Pain Interference With Subject's Sleep
Description: as for outcome 14
Time Frame: Baseline Week, Visit 6
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 162 | 161 | 163
units on a scale | -1.9 (2.15) | -2.0 (2.28) | -2.2 (2.26)

18. Secondary Outcome: Within-subject Change From the Baseline Week to Visit 7 in Daily Perception of Pain Interference With Subject's Sleep
Description: as for outcome 14
Time Frame: Baseline Week, Visit 7
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 157 | 151 | 151
units on a scale | -2.2 (2.19) | -2.3 (2.22) | -2.5 (2.37)

19. Secondary Outcome: Within-subject Change From the Baseline Week to Visit 8 in Daily Perception of Pain Interference With Subject's Sleep
Description: as for outcome 14
Time Frame: Baseline Week, Visit 8
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 152 | 149 | 149
units on a scale | -2.1 (2.28) | -2.5 (2.26) | -2.5 (2.38)

20. Secondary Outcome: Within-subject Change From the Baseline Week to the Titration Phase in Daily Perception of Pain Interference With Subject's Sleep
Description: An 11-point Likert scale was used to assess the subject's sleep. The subject rated how the pain had interfered with sleep over the past 12 hours, from 0 (no interference) to 10 (complete interference). A lower value on the scale indicates improvement in symptoms. A negative change value indicates improvement from Baseline. Baseline Week was defined as the average of pain interference scores at the last 7 days prior to Visit 2. The value reported below is calculated as a difference between the average of the titration phase and the average of the Baseline Week.
Time Frame: Titration Phase (4 weeks), compared to the Baseline Week
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 177 | 186 | 176
units on a scale | -1.0 (1.54) | -1.3 (1.62) | -1.3 (1.67)

21. Secondary Outcome: Within-subject Change From the Baseline Week to the Maintenance Phase in Daily Perception of Pain Interference With Subject's Sleep
Description: An 11-point Likert scale was used to assess the subject's sleep. The subject rated how the pain had interfered with sleep over the past 12 hours, from 0 (no interference) to 10 (complete interference). A lower value on the scale indicates improvement in symptoms. A negative change value indicates improvement from Baseline. Baseline Week was defined as the average of pain interference scores at the last 7 days prior to Visit 2. The value reported below is calculated as a difference between the average of the maintenance phase and the average of the Baseline Week.
Time Frame: Maintenance Phase (12 weeks), compared to the Baseline Week
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 162 | 161 | 163
units on a scale | -2.0 (2.15) | -2.2 (2.22) | -2.4 (2.24)

22. Secondary Outcome: Within-subject Change From the Baseline Week to the Treatment Phase in Daily Perception of Pain Interference With Subject's Sleep
Description: An 11-point Likert scale was used to assess the subject's sleep. The subject rated how the pain had interfered with sleep over the past 12 hours, from 0 (no interference) to 10 (complete interference). A negative value indicates improvement in symptoms. A lower value on the scale indicates improvement in symptoms. A negative change value indicates improvement from Baseline. Baseline Week was defined as the average of pain interference scores at the last 7 days prior to Visit 2. The value reported below is calculated as a difference between the average of the treatment phase and the average of the Baseline Week.
Time Frame: Treatment Phase (16 weeks), compared to the Baseline Week
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 177 | 186 | 176
units on a scale | -1.6 (1.94) | -1.8 (1.94) | -2.0 (2.04)

23. Secondary Outcome: Within-subject Change From the Baseline Week to the Last 4 Weeks of Maintenance Phase in Daily Perception of Pain Interference With Subject's Sleep
Description: An 11-point Likert scale was used to assess the subject's sleep. The subject rated how the pain had interfered with sleep over the past 12 hours, from 0 (no interference) to 10 (complete interference). A lower value on the scale indicates improvement in symptoms. A negative change value indicates improvement from Baseline. Baseline Week was defined as the average of pain interference scores at the last 7 days prior to Visit 2. The value reported below is calculated as a difference between the average of the last available 28 days of maintenance for participants completing the maintenance phase (or the last 28 days prior to discontinuation for participants who discontinued in the titration or maintenance phase) and the average of the Baseline week.
Time Frame: Last 4 weeks of Maintenance Phase, compared to the Baseline Week
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 177 | 186 | 176
units on a scale | -1.9 (2.30) | -2.1 (2.24) | -2.3 (2.37)

24. Secondary Outcome: Within-subject Change From the Baseline Week to Visit 3 in Daily Perception of Pain Interference With Subject's General Activity
Description: An 11-point Likert scale was used to assess the subject's general activity. The subject rated how the pain had interfered with general activity over the past 12 hours, from 0 (no interference) to 10 (complete interference). A negative value indicates improvement from Baseline.
Time Frame: Baseline Week, Visit 3
Population: Only subjects with available data for subject's pain interference with subject's general activity at the respective are included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 177 | 187 | 177
units on a scale | -0.6 (1.30) | -0.7 (1.26) | -0.7 (1.40)

25. Secondary Outcome: Within-subject Change From the Baseline Week to Visit 4 in Daily Perception of Pain Interference With Subject's General Activity
Description: as for outcome 24
Time Frame: Baseline Week, Visit 4
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 171 | 181 | 170
units on a scale | -1.0 (1.57) | -1.3 (1.70) | -1.3 (1.84)

26. Secondary Outcome: Within-subject Change From the Baseline Week to Visit 5 in Daily Perception of Pain Interference With Subject's General Activity
Description: as for outcome 24
Time Frame: Baseline Week, Visit 5
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 168 | 171 | 169
units on a scale | -1.4 (1.83) | -1.6 (2.01) | -1.8 (2.11)

27. Secondary Outcome: Within-subject Change From the Baseline Week to Visit 6 in Daily Perception of Pain Interference With Subject's General Activity
Description: as for outcome 24
Time Frame: Baseline Week, Visit 6
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 162 | 162 | 164
units on a scale | -1.9 (2.15) | -2.0 (2.12) | -2.1 (2.28)

28. Secondary Outcome: Within-subject Change From the Baseline Week to Visit 7 in Daily Perception of Pain Interference With Subject's General Activity
Description: as for outcome 24
Time Frame: Baseline Week, Visit 7
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 157 | 152 | 152
units on a scale | -2.2 (2.24) | -2.3 (2.11) | -2.3 (2.37)

29. Secondary Outcome: Within-subject Change From the Baseline Week to Visit 8 in Daily Perception of Pain Interference With Subject's General Activity
Description: as for outcome 24
Time Frame: Baseline Week, Visit 8
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 152 | 150 | 150
units on a scale | -2.1 (2.29) | -2.4 (2.15) | -2.4 (2.42)

30. Secondary Outcome: Within-subject Change From the Baseline Week to the Titration Phase in Daily Perception of Pain Interference With Subject's General Activity
Description: An 11-point Likert scale was used to assess the subject's general activity. The subject rated how the pain had interfered with general activity over the past 12 hours, from 0 (no interference) to 10 (complete interference). A negative value indicates improvement from Baseline. The value reported below is calculated as a difference between the average of the titration phase and the average of the Baseline Week.
Time Frame: Titration Phase (4 weeks), compared to the Baseline Week
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 177 | 187 | 177
units on a scale | -1.0 (1.50) | -1.2 (1.60) | -1.3 (1.72)

31. Secondary Outcome: Within-subject Change From the Baseline Week to the Maintenance Phase in Daily Perception of Pain Interference With Subject's General Activity
Description: An 11-point Likert scale was used to assess the subject's general activity. The subject rated how the pain had interfered with general activity over the past 12 hours, from 0 (no interference) to 10 (complete interference). A negative value indicates improvement from Baseline. The value reported below is calculated as a difference between the average of the maintenance phase and the average of the Baseline Week.
Time Frame: Maintenance Phase (12 weeks), compared to the Baseline Week
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 162 | 162 | 164
units on a scale | -2.0 (2.17) | -2.2 (2.05) | -2.2 (2.27)

32. Secondary Outcome: Within-subject Change From the Baseline Week to the Treatment Phase in Daily Perception of Pain Interference With Subject's General Activity
Description: An 11-point Likert scale was used to assess the subject's general activity. The subject rated how the pain had interfered with general activity over the past 12 hours, from 0 (no interference) to 10 (complete interference). A negative value indicates improvement from Baseline. The value reported below is calculated as a difference between the average of the treatment phase and the average of the Baseline Week.
Time Frame: Treatment Phase (16 weeks), compared to the Baseline Week
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 177 | 187 | 177
units on a scale | -1.6 (1.94) | -1.8 (1.85) | -1.9 (2.06)

33. Secondary Outcome: Within-subject Change From the Baseline Week to the Last 4 Weeks of the Maintenance Phase in Daily Perception of Pain Interference With Subject's General Activity
Description: An 11-point Likert scale was used to assess the subject's general activity. The subject rated how the pain had interfered with general activity over the past 12 hours, from 0 (no interference) to 10 (complete interference). A negative value indicates improvement from Baseline. The value reported below is calculated as a difference between the average of the last available 28 days of maintenance for participants completing the maintenance phase (or the last 28 days prior to discontinuation for participants who discontinued in the titration or maintenance phase) and the average of the Baseline week.
Time Frame: Last 4 weeks of Maintenance Phase, compared to the Baseline Week
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 177 | 187 | 177
units on a scale | -1.9 (2.30) | -2.1 (2.16) | -2.2 (2.38)

34. Secondary Outcome: Percentage of Days of Rescue Medication Use During the Treatment Phase
Description: Percentage of days of rescue medication use was the number of days in the visit/trial phase with rescue medication use divided by the total number of days in the visit/trial phase times 100.
Time Frame: During the Treatment Phase (up to 16 weeks)
Population: Only subjects with available data for rescue medication use are included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 177 | 188 | 177
percentage of days | 6.6 (20.27) | 7.0 (20.28) | 9.1 (23.67)

35. Secondary Outcome: Within-subject Change From Baseline to Visit 8 in Subject's Quality of Life
Description: Quality of life was analyzed using the Short Form-36 (SF-36) Health Survey. The SF-36 is a participant self-rated questionnaire which consists of 8 sub-scores ranging from 0-100 with higher scores indicating a better health state. The sub-scores are: 1. Physical Functioning, 2. Role-Physical, 3. Bodily Pain, 4. General Health, 5. Vitality, 6. Social Functioning, 7. Role-Emotional, 8. Mental Health. Items 1-4 contribute to the physical component Summary (PCS) score. Items 5-8 contribute to the mental component summary (MCS) score. The PCS and MCS were based on the standardized values of the 8 domains. The maximum and minimum possible values for PCS and MCS is 0-100, where higher scores indicate good condition. A positive change value indicates improvement from baseline. As pre-specified in SAP, values were planned to be summarized and disclosed by placebo and LCM 400 mg/day (pooled) groups.
Time Frame: Baseline, Visit 8
Population: A total of 177 subjects treated with Placebo and 365 subjects treated with lacosamide were initially included in the Full Analysis Set. Only subjects with available data for change from Baseline to Visit 8 in the sub-scores of subject's quality of life are included in the analysis. Number of subjects analyzed is given separately per sub-score.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lacosamide Pooled FT and ST: Subjects received LCM as Fast Titration (FT) or Standard Titration (ST).
Arm/Group | Placebo | Lacosamide Pooled FT and ST
Number analyzed (Participants) | 177 | 365
units on a scale
  Physical Functioning: number analyzed (Participants) | 169 | 345
  Physical Functioning | 3.8 (16.30) | 4.4 (18.85)
  Role-Physical: number analyzed (Participants) | 168 | 345
  Role-Physical | 15.3 (37.80) | 10.3 (39.33)
  Bodily Pain: number analyzed (Participants) | 169 | 345
  Bodily Pain | 13.4 (20.51) | 16.9 (19.99)
  General Health: number analyzed (Participants) | 169 | 343
  General Health | 5.0 (15.09) | 4.8 (15.39)
  Vitality: number analyzed (Participants) | 169 | 344
  Vitality | 4.4 (16.12) | 7.5 (17.94)
  Social Functioning: number analyzed (Participants) | 169 | 345
  Social Functioning | 8.4 (23.05) | 5.1 (22.37)
  Role-Emotional: number analyzed (Participants) | 168 | 345
  Role-Emotional | 6.5 (44.42) | 4.7 (47.28)
  Mental Health: number analyzed (Participants) | 169 | 344
  Mental Health | 3.5 (16.97) | 4.8 (18.60)
  PCS: number analyzed (Participants) | 168 | 342
  PCS | 3.9 (6.61) | 4.0 (6.99)
  MCS: number analyzed (Participants) | 168 | 342
  MCS | 1.9 (10.06) | 1.8 (10.91)

36. Secondary Outcome: Percentage of Patients With Categorized Patient's Global Impression of Change in Pain (PGIC) at Visit 8
Description: The PGIC is a 7-point categorical rating scale in which the subject rates the change in his/her pain since starting trial medication. Categories are as following: much worse, moderately worse, mildly worse, no change, mildly better, moderately better, much better. As pre-specified in SAP, values were planned to be summarized and disclosed by placebo and LCM 400 mg/day (pooled) reporting groups.
Time Frame: Visit 8
Population: Only subjects with available data for Patient's Global Impression of Change in Pain are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lacosamide Pooled FT and ST
Number analyzed (Participants) | 171 | 343
percentage of participants
  Much worse | 1.2 | 0.6
  Moderately worse | 1.2 | 1.7
  Mildly worse | 3.5 | 2.6
  No change | 23.4 | 17.8
  Mildly better | 31.6 | 23.3
  Moderately better | 26.9 | 32.4
  Much better | 12.3 | 21.6

37. Secondary Outcome: Percentage of Patients With Categorized Satisfaction With Medications at Visit 8
Description: Categories of satisfaction are as following: very satisfied, satisfied, neither satisfied/dissatisfied, dissatisfied, very dissatisfied, not applicable, not done (no data available).
Time Frame: Visit 8
Population: Only subjects with available data for satisfaction with medications are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 171 | 178 | 168
percentage of participants
  Very Satisfied | 11.7 | 14.0 | 15.5
  Satisfied | 43.9 | 45.5 | 50.0
  Neither Satisfied/Dissatisfied | 25.7 | 24.2 | 23.8
  Dissatisfied | 11.7 | 11.8 | 8.3
  Very Dissatisfied | 4.1 | 2.8 | 0.6
  Not Applicable | 0 | 0.6 | 0
  Not Done | 2.9 | 1.1 | 1.8

38. Secondary Outcome: Change From Baseline in Medical Outcomes Study (MOS) Sleep Scale Scores at Visit 8
Description: The MOS Sleep scale is used to assess the subject's quality of sleep. The scale consists of 12 individual items categorized into two sleep problems indices (SPI I/II) and 5 subscales: sleep disturbance, sleep somnolence, snoring, short of breath (SoB) or headache, sleep adequacy. Scores range from 0 to 100. Sleep adequacy scale: High values indicate a high quality of sleep. A positive change indicates improvement in quality of sleep. All other Sleep Scales: Low values indicate a high quality of sleep. A negative change indicates improvement in quality of sleep.
Time Frame: Baseline, Visit 8
Population: 177 subjects treated with Placebo, 188 subjects treated with Lacosamide FT and 177 subjects treated with Lacosamide ST were initially included in the FAS. Only subjects with available data for change from Baseline to Visit 8 in MOS sleep scale scores are included in the analysis. Number of subjects analyzed is given separately per sub-score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lacosamide FT | Lacosamide ST
Number analyzed (Participants) | 177 | 188 | 177
units on a scale
  Sleep Disturbance: number analyzed (Participants) | 105 | 116 | 106
  Sleep Disturbance | -13.4 (19.30) | -15.2 (22.65) | -17.1 (23.97)
  Sleep Somnolence: number analyzed (Participants) | 105 | 116 | 106
  Sleep Somnolence | -7.0 (16.25) | -2.1 (19.69) | -4.6 (20.41)
  Snoring: number analyzed (Participants) | 105 | 115 | 104
  Snoring | -2.7 (27.33) | 0.0 (25.13) | -6.7 (27.25)
  SoB/ Headache: number analyzed (Participants) | 105 | 116 | 106
  SoB/ Headache | -6.7 (23.32) | -1.0 (26.75) | -7.5 (24.76)
  Sleep Adequacy: number analyzed (Participants) | 105 | 116 | 106
  Sleep Adequacy | 7.2 (26.11) | 10.3 (26.37) | 15.1 (30.28)
  SPI I: number analyzed (Participants) | 105 | 116 | 106
  SPI I | -10.3 (15.15) | -8.3 (17.39) | -12.2 (19.58)
  SPI II: number analyzed (Participants) | 105 | 116 | 106
  SPI II | -10.6 (14.18) | -9.9 (16.66) | -13.1 (19.17)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline until the end of the trial (up to Week 18)
Description: Adverse Events refer to the Safety Set, consisting of all randomized subjects who took at least one dose of study medication. It was pre-specified in the Statistical Analysis Plan that AEs will be summarized and disclosed for placebo and LCM 400 mg/day (pooled) for all participants, who took at least one dose of medication (Safety Set). AEs were planned to be collected and summarized irrespective of dosing strategy.
Arm/Group | Placebo | Lacosamide Pooled FT and ST
All-Cause Mortality (participants affected / at risk) | 0/179 | 0/370
Serious Adverse Events (participants affected / at risk) | 14/179 | 28/370
Other Adverse Events (participants affected / at risk) | 21/179 | 82/370
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=179) | Lacosamide Pooled FT and ST (N=370)
Atrial flutter (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Bundle branch block left (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Diabetic retinopathy (Eye disorders) | 1 | 0
Jejunitis (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Electrocardiogram PR prolongation (Investigations) | 1 | 0
Diabetic foot (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Toe deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Gastrinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1
Cerebellar syndrome (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Neuropathy (Nervous system disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 2
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Intestinal operation (Surgical and medical procedures) | 0 | 1
Arterial occlusive disease (Vascular disorders) | 0 | 2
Peripheral ischaemia (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=179) | Lacosamide Pooled FT and ST (N=370)
Vertigo (Ear and labyrinth disorders) | 2 | 21
Nausea (Gastrointestinal disorders) | 4 | 28
Nasopharyngitis (Infections and infestations) | 11 | 20
Dizziness (Nervous system disorders) | 3 | 29
Headache (Nervous system disorders) | 6 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days